CLINICAL TRIAL: NCT01803347
Title: Multicentre,Randomized,Comparative,Add-on,Into Two Parallel Groups Clinical Trial to Evaluate Efficacy and Safety of Autologous Mesenchymal Stem Cells Derived From Expanded Adipose Tissue (ASC), for Treatment of Complex Perianal Fistulizing Disease in Patients Without IBD.
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Stem Cells
Acronym: FISPAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-001178-28
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2017-03

CONDITIONS: Anal Fistula
Keywords: phase III; Adipose derived stem cells; Anal fistula; Cell therapy; Stem cell therapy
MeSH Terms: conditions — Rectal Fistula | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASC + fibrin glue (Experimental): Intervention: drug: ASC + fibrin glue Experimental: ASCs+fibrin glue: Subjects will be treated with a dose of 100 million ASCs plus fibrin glue plus a deep curettage and closure of the internal orifice and evaluated after 16 weeks. If needed a second dose of 100 million ASCs plus fibrin glue will be applied then.
  Interventions: Drug: ◦Drug: ASCs. + fibrin glue
- Fibrin glue (Active Comparator): Intervention: fibrin glue Fibrin glue: Subjects will be treated with a dose fibrin glue plus a deep curettage and closure of the internal orifice, and evaluated after 16 weeks. If needed a second dose of fibrin glue will be applied then.
  Interventions: Drug: fibrin glue

INTERVENTIONS:
Drug: ◦Drug: ASCs. + fibrin glue — Experimental group
  Other Names: Experimental Drug: ASCs + fibrin glue
  Arms: ASC + fibrin glue
Drug: fibrin glue — •Active Comparator: Fibrin glue Intervention: Drug: Fibrin adhesive
  Arms: Fibrin glue

SUMMARY:
Efficacy of treatment of perianal fistula with mesenchymal stem cells and surgery

DETAILED DESCRIPTION:
Study of efficacy of adipose derived mesenchimals stem cells and surgery to treat complex perianal fistula

ELIGIBILITY:
Inclusion Criteria:

1. Signature of informed consent.
2. Complex perianal fistula cryptoglandular. Understood as a fistula in which at least one of the following circumstances is present:

   * some degree of fecal incontinence associated
   * extrasphinterics fistulas,
   * fistulas supraresfinterianas
   * high transsphincteric fistulas.
3. Patients of both genders, with more that 18 years.
4. Good overall health, according to data from the clinical history and physical examination.

Exclusion Criteria:

1. Patient diagnosed with inflammatory bowel disease.
2. Subjects with abscess, except if a complete cleaning of the drainage area of collections is performed and the absence of abscess and other collections larger than 2 cm in maximum diameter before treatment is started is confirmed.
3. History of alcohol or substance abuse in the 6 months prior to inclusion.
4. Malignancy, except in the case of basal cell carcinoma or squamous cell skin or a history of malignancy, unless they have been found in remission during the previous 5 years.
5. medical or psychiatric illness of any kind which, in the opinion of the investigator, may be a reason for exclusion from the study.
6. Subjects with congenital or acquired immunodeficiencies. Treponema, Hepatitis B and / or C or tuberculosis diagnosed at the time of inclusion.
7. Major surgery or severe trauma of the subject in the previous semester.
8. Pregnant or lactating women.
9. Adult women of childbearing potential not using effective contraception during the trial.
10. Administration of any investigational drug at present to three months prior to enrollment for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Safety/efficacy | 2014, march
  Closure of fistulas defined as absence of suppuration and re-epithelization of the external opening and absence of collections>2 cm directly related to the fistula tract treated, as measured by MRI (healing) [ Time Frame: weeks 1, 4, 12 and 16. Week 28 in patients with a second dose ]

SECONDARY OUTCOMES:
Safety/efficacy | 2015, march
  Clinical complexity of fistula (complexity of fistula score) • Safety: Cumulative incidence of adverse effects. • Quality of life (SF-36 score) • Degree of anal incontinence (Wexner incontinence score) [ Time Frame: weeks 1, 4, 12 and 16. Week 28 in patients with a second dose ]

CONTACTS AND LOCATIONS:
Overall Officials: Damián García-Olmo, Prof., Principal Investigator — Instituto de Investigación Hospital Universitario La Paz
Locations (5):
- Spain (5):
  - Hospital Clínico Lozano Blesa, Zaragoza, Aragon
  - Hospital Clínico Universitario, Salamanca, Castille and León
  - Hospital General Universitario, Valencia, Valencia
  - Hospital Universitario La Paz, Madrid
  - Clínica Universitaria de Navarra, Pamplona

REFERENCES:
- [Result] de la Portilla F, Alba F, Garcia-Olmo D, Herrerias JM, Gonzalez FX, Galindo A. Expanded allogeneic adipose-derived stem cells (eASCs) for the treatment of complex perianal fistula in Crohn's disease: results from a multicenter phase I/IIa clinical trial. Int J Colorectal Dis. 2013 Mar;28(3):313-23. doi: 10.1007/s00384-012-1581-9. Epub 2012 Sep 29. PMID 23053677
- [Result] Guadalajara H, Herreros D, De-La-Quintana P, Trebol J, Garcia-Arranz M, Garcia-Olmo D. Long-term follow-up of patients undergoing adipose-derived adult stem cell administration to treat complex perianal fistulas. Int J Colorectal Dis. 2012 May;27(5):595-600. doi: 10.1007/s00384-011-1350-1. Epub 2011 Nov 9. PMID 22065114
- [Result] Garcia-Arranz M, Gomez-Pinedo U, Hardisson D, Herreros D, Guadalajara H, Garcia-Gomez I, Garcia-Verdugo JM, Garcia-Olmo D. Histopathological analysis of human specimens removed from the injection area of expanded adipose-derived stem cells. Histopathology. 2010 Jun;56(7):979-82. doi: 10.1111/j.1365-2559.2010.03573.x. No abstract available. PMID 20636801
- [Result] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Result] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359
- [Result] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795